CLINICAL TRIAL: NCT00133250
Title: Value of Abciximab in Patients With AMI Undergoing PCI After High Dose Clopidogrel Pretreatment (BRAVE 3)
Brief Title: Value of Abciximab in Patients With AMI Undergoing Primary PCI After Clopidogrel Pretreatment (BRAVE 3)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. I00902
Record Dates: First submitted 2005-08-20; First posted 2005-08-23 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Abciximab
  Interventions: Drug: Abciximab
- B (Placebo Comparator): Heparin Sodium
  Interventions: Other: Placebo Heparin Sodium

INTERVENTIONS:
Drug: Abciximab — Abciximab bolus and infusion is given. Study medication includes 3 identical vials, each with 5 ml solution containing 10 mg abciximab. The bolus dose to be given should be rated at 0.125 ml/kg of patient's weight. After the bolus, a total dose of 0.045 ml/kg study substance (up to a maximal quantity of 3.6 ml) should be given over 12 hours.
  Other Names: ReoPro
  Arms: A
Other: Placebo Heparin Sodium — Placebo bolus plus infusion is given. Study medication includes 3 identical vials, each with 5 ml solution containing 3000 U Heparin. The bolus dose to be given should be rated at 0.125 ml/kg of patient's weight. After the bolus, a total dose of 0.045 ml/kg study substance (up to a maximal quantity of 3.6 ml) should be given over 12 hours.
  Arms: B

SUMMARY:
The purpose of this study is to assess whether abciximab is associated with additional benefit in patients with AMI treated with PCI after high dose clopidogrel loading.

DETAILED DESCRIPTION:
The goal of all reperfusion therapies in acute myocardial infarction (AMI) is an effective restoration of coronary blood flow and the reduction of infarct size. Recently, the researchers were able to achieve excellent results with primary stenting plus abciximab in terms of reduction of infarct size and improvement of clinical outcome in the STOPAMI trial. This strategy provided a clear benefit compared to fibrinolysis. On the basis of the data published in the last 2 years, hospitals without angioplasty facilities have now better possibilities to improve the results of primary treatment of patients with AMI by immediately referring these patients to highly experienced centers in coronary interventions. There is an increasing interest to assess the additional advantages of pharmacologic reperfusion approaches which are readily applicable in the time window between presentation and arrival at the catheterization room. Two studies have shown that the results of the PCI in patients with AMI pretreated with fibrinolysis may even be more unfavorable than those achieved with angioplasty alone. Glycoprotein (GP) IIb/IIIa blocker abciximab has been shown to improve the results of the primary PCI in AMI. However, no rapidly effective antiplatelets therapy was available at the time when the studies on the benefit of abciximab were performed. Recent studies have shown that a high, 600 mg loading dose of clopidogrel is significantly more rapidly acting and that maximal inhibition of platelet aggregation is achieved within 2 hours after administration. In the ISAR-REACT trial, a high loading dose of clopidogrel was well tolerated, associated with such a low frequency of procedural complications that the use of abciximab offered no clinically measurable benefit at 30 days.

Comparison:

Abciximab (bolus+infusion for 12h) versus Placebo (bolus+infusion for 12h) after pre-treatment with 600 mg clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with ST-Elevation acute myocardial infarction within 24 hours from the onset of symptoms

Exclusion Criteria:

* Age >80 years
* Malignancies
* Cardiogenic shock
* Prolonged cardio-pulmonary resuscitation
* Increased risk of bleeding
* Relevant hematologic deviations (hemoglobin <100 g/L or hematocrit <34%, platelet count <100 x 10^9 /L or platelet count >600 x 10^9 /L)
* Known allergy to the study medication
* Pregnancy (present or suspected)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2003-06; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular infarct size calculated as the final perfusion defect at follow-up scintigraphic study | 5-7 days

SECONDARY OUTCOMES:
Clinical adverse events (death of any cause, reinfarction, stroke, urgent reinterventions, major and minor bleeding complications, thrombocytopenia <20 x 10^9 /L) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (5):
- Allgemeines Krankenhaus Wien, Vienna, Austria
- Germany (4):
  - Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - Deutsches Herzzentrum Muenchen, Munich
  - First Medizinische Klinik, Klinikum rechts der Isar, Munich
  - Klinikum Traunstein, Traunstein

REFERENCES:
- [Background] Weaver WD, Simes RJ, Betriu A, Grines CL, Zijlstra F, Garcia E, Grinfeld L, Gibbons RJ, Ribeiro EE, DeWood MA, Ribichini F. Comparison of primary coronary angioplasty and intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review. JAMA. 1997 Dec 17;278(23):2093-8. PMID 9403425
- [Background] Vermeer F, Oude Ophuis AJ, vd Berg EJ, Brunninkhuis LG, Werter CJ, Boehmer AG, Lousberg AH, Dassen WR, Bar FW. Prospective randomised comparison between thrombolysis, rescue PTCA, and primary PTCA in patients with extensive myocardial infarction admitted to a hospital without PTCA facilities: a safety and feasibility study. Heart. 1999 Oct;82(4):426-31. doi: 10.1136/hrt.82.4.426. PMID 10490554
- [Background] Neumann FJ, Blasini R, Schmitt C, Alt E, Dirschinger J, Gawaz M, Kastrati A, Schomig A. Effect of glycoprotein IIb/IIIa receptor blockade on recovery of coronary flow and left ventricular function after the placement of coronary-artery stents in acute myocardial infarction. Circulation. 1998 Dec 15;98(24):2695-701. doi: 10.1161/01.cir.98.24.2695. PMID 9851955
- [Background] Muller I, Seyfarth M, Rudiger S, Wolf B, Pogatsa-Murray G, Schomig A, Gawaz M. Effect of a high loading dose of clopidogrel on platelet function in patients undergoing coronary stent placement. Heart. 2001 Jan;85(1):92-3. doi: 10.1136/heart.85.1.92. No abstract available. PMID 11119474
- [Background] Kastrati A, Mehilli J, Schlotterbeck K, Dotzer F, Dirschinger J, Schmitt C, Nekolla SG, Seyfarth M, Martinoff S, Markwardt C, Clermont G, Gerbig HW, Leiss J, Schwaiger M, Schomig A; Bavarian Reperfusion Alternatives Evaluation (BRAVE) Study Investigators. Early administration of reteplase plus abciximab vs abciximab alone in patients with acute myocardial infarction referred for percutaneous coronary intervention: a randomized controlled trial. JAMA. 2004 Feb 25;291(8):947-54. doi: 10.1001/jama.291.8.947. PMID 14982910
- [Background] Kastrati A, Mehilli J, Schuhlen H, Dirschinger J, Dotzer F, ten Berg JM, Neumann FJ, Bollwein H, Volmer C, Gawaz M, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment Study Investigators. A clinical trial of abciximab in elective percutaneous coronary intervention after pretreatment with clopidogrel. N Engl J Med. 2004 Jan 15;350(3):232-8. doi: 10.1056/NEJMoa031859. PMID 14724302
- [Background] Kastrati A, Mehilli J, Dirschinger J, Schricke U, Neverve J, Pache J, Martinoff S, Neumann FJ, Nekolla S, Blasini R, Seyfarth M, Schwaiger M, Schomig A; Stent versus Thrombolysis for Occluded Coronary Arteries in Patients With Acute Myocardial Infarction (STOPAMI-2) Study. Myocardial salvage after coronary stenting plus abciximab versus fibrinolysis plus abciximab in patients with acute myocardial infarction: a randomised trial. Lancet. 2002 Mar 16;359(9310):920-5. doi: 10.1016/S0140-6736(02)08022-4. PMID 11918909
- [Result] Mehilli J, Kastrati A, Schulz S, Frungel S, Nekolla SG, Moshage W, Dotzer F, Huber K, Pache J, Dirschinger J, Seyfarth M, Martinoff S, Schwaiger M, Schomig A; Bavarian Reperfusion Alternatives Evaluation-3 (BRAVE-3) Study Investigators. Abciximab in patients with acute ST-segment-elevation myocardial infarction undergoing primary percutaneous coronary intervention after clopidogrel loading: a randomized double-blind trial. Circulation. 2009 Apr 14;119(14):1933-40. doi: 10.1161/CIRCULATIONAHA.108.818617. Epub 2009 Mar 30. PMID 19332467
- [Derived] Schulz S, Birkmeier KA, Ndrepepa G, Moshage W, Dotzer F, Huber K, Dirschinger J, Seyfarth M, Schomig A, Kastrati A, Mehilli J. One-year clinical outcomes with abciximab in acute myocardial infarction: results of the BRAVE-3 randomized trial. Clin Res Cardiol. 2010 Dec;99(12):795-802. doi: 10.1007/s00392-010-0185-z. Epub 2010 Jun 27. PMID 20582594